CLINICAL TRIAL: NCT06006247
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of CVN424 in Early Parkinson's Disease
Brief Title: Early Parkinson's Disease Monotherapy With CVN424
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerevance Beta, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cerevance (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVN424-203
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; CVN424; Progressive neurodegenerative disorder; Parkinson's disease monotherapy
MeSH Terms: conditions — Parkinson Disease; Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CVN424 150 mg (Experimental): Participants will be administered with CVN424 150 mg.
  Interventions: Drug: CVN424 150 mg
- Placebo (Placebo Comparator): Participants will be administered with placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CVN424 150 mg — Participants will receive 1 CVN424 tablet (150 mg) per day.
  Arms: CVN424 150 mg
Drug: Placebo — Participants will receive 1 matching placebo tablet per day.
  Arms: Placebo

SUMMARY:
This is a multicenter, 12-week, placebo-controlled clinical trial of CVN424 150 milligrams (mg) tablets in early, untreated Parkinson's Disease (PD). Participants will be randomized in a 1:1 ratio to CVN424 150 mg or placebo at the Baseline Visit. The purpose of this study is to measure effect on motor features with CVN424 tablets compared to placebo in early, untreated PD and to evaluate the potential of CVN424 to improve motor and non-motor functions in participants with early PD who are not taking dopaminergic or anti-PD therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD consistent with United Kingdom Brain Bank and Movement Disorder Society Research Criteria for the Diagnosis of PD; must include bradykinesia with sequence effect, and motor asymmetry if no PD-type rest tremor.
* Not receiving anti-parkinsonian therapy, and not expecting to require it for the duration of the study.
* Men or women of all races who are at least 30 years at Screening.
* Modified Hoehn and Yahr ≤ 2.5 at Screening.
* Montreal Cognitive Assessment (MoCA) ≥ 26.
* Freely ambulatory at time of Screening (with/without assistive device).
* Female participants of childbearing potential and male participants with female partners of childbearing potential must agree to either remain abstinent or use adequate and reliable contraception throughout the study and at least 30 days after the last dose of study drug has been taken.
* Able and willing to give written (signed and dated) informed consent approved by an institutional review board, and to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures to complete the study.
* Approved as an appropriate and suitable candidate by the Enrollment Authorization Committee (EAC).

Exclusion Criteria:

* Diagnosis of secondary or atypical parkinsonism.
* Diagnosis of parkinsonian motor signs or symptoms ≥ 4 years before Screening Visit.
* Previous surgical procedure for PD.
* Prior treatment with a dopamine agonist, levodopa, monoamine oxidase B (MAOB) inhibitor, or adenosine A2A receptor antagonists for more than 28 total days prior to screening. Additional exclusionary parameters around PD treatment include:
* Treatment with a dopamine agonist within 14 days of Screening.
* Treatment with a MAOB inhibitor within 90 days of Screening.
* Current use of any antipsychotic, metoclopramide, or reserpine. If previously used, this may not have been within 28 days of Screening or 5 elimination half-lives (whichever one is longer).
* Current use of potent Cytochrome P450 (CYP) 3A4/5 inhibitors or inducers.
* Clinically significant orthostatic hypotension.
* Clinically significant hallucinations requiring antipsychotic use.
* Known autoimmune, malignancy (except basal cell carcinoma) or hematologic disease (prior or current) likely to interfere with the safe participation of the participant or interfere with assessment of safety or efficacy based on the opinion of the investigator and the medical monitor.
* Any clinically significant medical, surgical, or psychiatric abnormality that, in the judgment of the Investigator, is likely to interfere with study compliance, the safe participation of the participant or the assessment of safety or efficacy.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 2 times the upper limit of normal (ULN), and total bilirubin greater than 1.5 times ULN.
* Participants with Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided that direct bilirubin is ≤ 1.5 times ULN.
* Significant renal impairment as determined by estimated glomerular filtration rate (eGFR) using creatinine clearance (CrCL) as per the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of ≤ 50 milliliters per minutes (mL/min).
* Participant has an ECG, prior documentation history, or clinical evidence of potentially unstable heart disease, including, but not limited to the following:

  1. QT interval corrected using Fridericia's formula (QTcF) > 470 milliseconds (msec) for female participants; > 450 msec for male participants
  2. Complete right or left bundle branch block
  3. Myocardial infarction within 1 year prior to screening, unstable angina within 6 months, or a current concern for symptomatic ischemic heart disease in the opinion of the investigator
  4. Clinically significant atrial or ventricular dysrhythmia; the heart must be in predominantly normal sinus rhythm
  5. Second- or third-degree atrioventricular (AV) block
  6. New York Heart Association (NYHA) Class II or higher congestive heart failure
  7. Clinically significant cardiomyopathy or cardiac structural abnormality, in the opinion of the investigator
  8. Any other cardiac condition that the Investigator feels may predispose the participant to ischemia or arrhythmia
* Current (or within past 12 months) diagnosis or history of substance abuse (excluding nicotine or caffeine) by Diagnostic and Statistical Manual of Mental Disorders 5 criteria.
* Positive urine drug screen for tetrahydrocannabinol or any drugs that may affect participant safety or interfere with efficacy assessments.
* Medical or recreational use of marijuana within 2 months of the Screening Visit. Use of cannabidiol (CBD) is prohibited after the Screening Visit and throughout the study.
* Currently active major depression as determined by Beck Depression Inventory (BDI)-II score of > 19.
* Active suicidal ideation within 1 year prior to Screening Visit as determined by a positive response to Question 4 or 5 on the C-SSRS.
* Currently lactating or pregnant, or planning to become pregnant during the study.
* Current participation in another investigational clinical study and/or receipt of any investigational drug within 90 days prior to Screening.
* Prior use of CVN424 investigational product.
* Positive test for coronavirus disease 2019 (COVID-19). A participant who tests positive for COVID-19 will be eligible to be rescreened once result is negative.
* Positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) consistent with current infection.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 on the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II + Part III | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same approved rater throughout the study. Part II scores motor aspects of experiences of daily living based on 13 items, it is a self-administered questionnaire completed by the participant, which can be reviewed by the Investigator to ensure all responses are completed. Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0 (normal) to 4(severe). A 0 means there is no disability, and the higher the score, the more the disability is reflected. The maximum score for Part III is 132. The total score is the sum of the numerical response values of the items. It is completed by a rater based on findings from the motor examination.

SECONDARY OUTCOMES:
Change from Baseline to Week 12 on the MDS-UPDRS Part III | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same clinician throughout the study. Part III consists of 33 scores based on 18 items, and each question is anchored with five response scale from 0 (normal) to 4(severe). A 0 means there is no disability, and the higher the score, the more the disability is reflected. The maximum score for Part III is 132. The total score is the sum of the numerical response values of the items. It is completed by a rater based on findings from the motor examination.
Change from Baseline to Week 12 on the Clinical Global Impression Scale - Severity (CGI-S) | Baseline and Up to Week 12
  The CGI-S is a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal/not at all ill) to 7 (amongst the most severely ill participants). This requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. Higher scores indicate worser the illness.
Change from Baseline to Week 12 on the Patient Global Impression Scale - Severity (PGI-S) | Baseline and Up to Week 12
  The PGI-S is a participant-completed assessment rating PD severity on a scale of 1 to 5 with 1 being none and 5 being very severe. Higher scores indicate worser the illness.
Change from Baseline to Week 12 on the MDS-UPDRS Part II | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same clinician throughout the study. Part II assess motor experiences of daily living, motor aspects of experiences of daily living. This part has 13 items. It is a self-administered questionnaire completed by the participant, which can be reviewed by the Investigator to ensure all responses are completed.
Change from Baseline to Week 12 on the MDS-UPDRS Part I | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same clinician throughout the study. Part I assess non-motor experiences of daily living, non-motor aspects of experiences of daily living (6 items assessed by interview and 7 items by self-assessment). It has 13 items and is further grouped into two parts: Part IA has items associated with behaviors that are assessed and completed by the rater based on information provided by the participant and caregiver. Part IB is self-administered and completed by the participant with or without assistance or input from the caregiver, but independently of the rater. Responses to both IA and IB can be reviewed by the rater to ensure information accuracy and/or provide additional information or clarification of the test items, if necessary.
Change from Baseline on the Epworth Sleepiness Scale (ESS) | Baseline and Up to Week 12
  The ESS is a participant self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0 to 3: would never doze, slight chance of dozing, moderate chance of dozing, and high chance of dozing), their usual chances of dozing off or falling asleep while engaged in eight different activities, such as sitting and reading, watching television, sitting in a public place, etc. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their "daytime sleepiness". The questionnaire takes no more than 2 or 3 minutes to answer.
Change from Baseline on the Non-motor Symptoms Scale (NMSS) | Baseline and Up to Week 12
  The NMSS for Parkinson's Disease is a 30-item rater-based scale to assess the frequency and severity of NMSS in participants across all stages of PD. The NMSS measures the severity and frequency of non-motor symptoms across 9 dimensions (cardiovascular, including falls, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastrointestinal, urinary, sexual function, and miscellany). Responses are to quantify symptoms according to severity (using a scale of 0 to 3) and frequency (using a scale of 0 to 4). It is completed by a rater.
Change from Baseline on the total MDS-UPDRS | Baseline and Up to Week 12
  The MDS-UPDRS is a comprehensive 50-question assessment of both motor and non-motor symptoms associated with PD. It features sections that require independent completion by people with PD and their caregivers, and sections to be completed by the same clinician throughout the study. The total score of MDS-UPDRS is the sum of Parts I, II and III.
Change from Baseline on the Parkinson's Disease Sleep Scale (PDSS-2) | Baseline and Up to Week 12
  The PDSS-2 is a 15-item participant-reported outcome measure to assess nocturnal disturbances in PD. It is a 5-point frequency scale (from "very often" [0] to "never" [4]), with a total score ranging from 0 to 60, where higher scores indicate greater impairment.
Number of participants reporting treatment emergent adverse events (TEAEs), TEAEs related to moderate or severe intensity and leading to withdrawal of study drug | Up to Week 14
Number of participants reporting serious adverse events (SAEs) | Up to Week 14
Number of participants with clinically significant changes in physical examination, vital signs, electrocardiogram (ECG) finding, laboratory values and Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Week 14
Number of participants reporting abuse related adverse events | Up to Week 14
Number of participants with occurrences of withdrawal symptoms recorded at the follow-up visit | At Week 14
Percentage of completers | Up to Week 14

OTHER OUTCOMES:
Change from Baseline to Week 12 on the Modality Virtual Assessment | Baseline and Up to Week 12
  The Modality System is an artificial intelligence interface designed to collect information on clinical performance through audio-visual conversational technology. Participants will engage with a virtual agent via a web browser on their electronic device, completing assessments aimed at testing various functions including speech, visuo-motor skills, prosodic (stress and intonation patterns), cognitive, and linguistic abilities.
Change from Baseline to Week 12 on the CogState digital cognitive battery | Baseline and Up to Week 12
  Cogstate Digital Cognitive Testing Battery are computerized cognitive assessments of attention, executive function, verbal learning, and memory. It uses standardized scores to assess participant's cognitive function. These scores are transformed into a scale where the average performance of the general population is set at 100, with a standard deviation of 15. This means that a score of 100 represents average cognitive function, while scores above or below indicate better or poorer performance, respectively, compared to the average.
Change from Baseline to Week 12 on the Schwab and England Activities of Daily Living (ADL) | Baseline and Up to Week 12
  The Schwab and England (S & E) Activities of Daily Living (ADL) Scale is a commonly used tool to measure daily function for Parkinson's disease (PD). The S & E Scale rates a PD participant's function on a scale from 0 indicating worst possible function to 100 indicating no impairment.
Change from Baseline to Week 12 on the Starkstein Apathy Scale (SAS) | Baseline and Up to Week 12
  The SAS instrument is used to identify apathy in participants with PD. The scale comprises 14 questions in which the respondent self-rates on a 4-point scale, ranging from "Not at all", "Slightly", "Some", and "A Lot". Ratings are a score from 3 to 0 for questions 1-8, and from 0 to 3 for questions 9-14, producing a total score out of 42. A score above 14 is considered the more severe level of apathy.
Change from Baseline to Week 12 on the Electroencephalogram (EEG) derived sleep metrics | Baseline and Up to Week 12
  Beacon Dreem overnight EEG is a wearable device that will collect EEG signals to measure sleep patterns and quality. Data will be collected for 3 consecutive nights before or after specified in-person clinic visits.
Change from Baseline to Week 12 on the Parkinson's Disease Patient Report of Problems (PD-PROP™) | Baseline and Up to Week 12
  The PD-PROP™ is a questionnaire with open-ended questions that asks individuals with PD to rank, in their own words, without restriction of content or length, up to 5 PD-related bothersome problems and their related effects on daily functioning.
Change from Baseline to Week 12 on the Personal Wellbeing Patient Report of Problems (PWB-PROP™) | Baseline and Up to Week 12
  The PWB-PROP™ is a questionnaire with open-ended questions that asks individuals with PD to rank, in their own words, without restriction of content or length, up to 5 PD-related bothersome problems related to their day-to-day life or personal wellbeing, such as personal, family, financial, social, or other aspects and their related effects on daily functioning.
Change from Plasma concentration of CVN424 | Pre-dose (0 h) and at 4 h post-dose on Day 1, Week 4, 8, and 12
  Blood samples will be collected at various timepoints for analysis of plasma concentration of CVN424.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - St Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Muhammad Ali Parkinson Center, Phoenix, Arizona
  - Movement Disorders Center of Arizona, LLC, Scottsdale, Arizona
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - N1 Research LLC, Orlando, Florida
  - Parkinson's Disease Treatment Center of SWFL, Port Charlotte, Florida
  - University of South Florida Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Dept of Neurology Kentucky Neuroscience Institute Research, Lexington, Kentucky
  - University of Kentucky, Center for Clinical and Translational Sciences, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Hospital / Michigan Clinical Research Unit (MCRU) Cardiovascular Center, Ann Arbor, Michigan
  - University of Michigan Department of Neurology, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Albany Medical Center, Albany, New York
  - Parkinson's Research Centers of America - Long Island, Commack, New York
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Riverhills Healthcare, Inc dba Riverhills Neuroscience, Cincinnati, Ohio
  - The Ohio State University Department of Neurology - Madden Center for Parkinson Disease and Other Movement Disorders, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Veracity Neuroscience, Memphis, Tennessee
  - Horizon Clinical Research Group, Cypress, Texas
  - Texas Movement Disorder Specialists, PLLC, Georgetown, Texas
  - Gill Neuroscience, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Inova Neurology - Fairfax, Fairfax, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - EvergreenHealth Neuroscience Institute, Kirkland, Washington
  - EvergreenHealth Research Department, Kirkland, Washington
  - Froedtert Hospital Department of Neurology, Milwaukee, Wisconsin
  - Medical College of Wisconsin Department of Neurology, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No